CLINICAL TRIAL: NCT04262141
Title: Investigator-Initiated Trial of the LSD1 Inhibitor IMG-7289 for the Treatment of Patients With Essential Thrombocythemia (ET) or Polycythemia Vera (PV) That Have Failed at Least One Standard Therapy
Brief Title: IMG-7289 in Patients With Essential Thrombocythemia (ET) or Polycythemia Vera (PV)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Terrence J Bradley, MD (Other)
Collaborators: Imago BioSciences, Inc., a subsidiary of Merck & Co., Inc., (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor-Investigator, Terrence J Bradley, MD, Assistant Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190932
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Essential Thrombocythemia; Polycythemia Vera
MeSH Terms: conditions — Thrombocythemia, Essential; Polycythemia Vera | interventions — bomedemstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMG-7289 in ET and PV Patients (Experimental): Oral daily dose of 0.6 mg/kg/day IMG-7289 will be administered:
  * The initial pilot period will enroll 8 participants to receive oral daily dose of IMG-7829 for 24 weeks, iteratively as long as there is clinical benefit in the absence of excess toxicity.
  * The second stage group will enroll an additional 16 participants to receive IMG-7829 for over 2 years, iteratively as long as there is clinical benefit in the absence of toxicity.
  Interventions: Drug: IMG-7289

INTERVENTIONS:
Drug: IMG-7289 — Daily oral dose of 0.6 mg/kg/day IMG-7829 capsules. Dose escalation an de-escalation rules applied as necessary.
  Other Names: IMG7289; IMG 7289

SUMMARY:
The purpose of this study is to assess the hematologic effects of IMG-7289 therapy in ET and PV patients who require platelet, White Blood Cell (WBC) or Red Blood Cell (RBC) control, and have failed at least one standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Diagnosis of Essential Thrombocythemia or Polycythemia Vera per World Health Organization (WHO) diagnostic criteria for myeloproliferative neoplasms (Arber et al., 2016).
3. Patients that have failed at least one standard therapy (failure is the equivalent of inadequate response or intolerance).
4. Platelet count >400 x 10^9/L pre-dose Day 1for patients with essential thrombocytopenia.
5. Platelet count >150 x 10^9/L pre-dose Day 1 for patients with polycythemia vera.
6. Peripheral blast count < 10% pre-dose Day 1.
7. Absolute neutrophil count (ANC) ≥ 0.5 x 10^9/L pre-dose Day 1.
8. Fibrosis score ≤ grade 2, as per a slightly modified version (Arber et al., 2016) of the European Consensus Criteria for Grading Myelofibrosis, (Thiele et al., 2005).
9. Life expectancy > 36 weeks.
10. Able to swallow capsules.
11. Amenable to blood draws, spleen size determination, bone marrow evaluations, and peripheral blood sampling during the study.
12. Must have discontinued prior therapy for condition under study for 2 weeks (4 weeks for interferon) prior to study drug initiation.
13. Agrees to use an approved method of contraception from Screening until 28 days after last administration of the study drug.
14. If male, agrees not to donate sperm or father a child for at least one month after the last dose of the study medication.

Exclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) questionnaire score of 3 or greater.
2. Currently pregnant, planning on being pregnant in the following 6 months or currently breastfeeding.
3. Currently residing outside the United States.
4. History of splenectomy.
5. Unresolved treatment related toxicities from prior therapies (unless resolved to ≤ Grade 1).
6. Uncontrolled active infection.
7. Known positive for HIV if not well-controlled (i.e., undetectable viral load), or infectious hepatitis, type A, B or C.
8. Current use of monoamine oxidase A and B inhibitors (MAOIs).
9. Evidence at the time of screening of increased risk of bleeding, including any of the following:

   * Activated partial thromboplastin time (aPTT) > 1.3 x the upper limit of normal
   * International normalized ratio (INR) >1.3 x the local upper limit of normal
   * History of severe thrombocytopenia or platelet dysfunction unrelated to a myeloproliferative disorder or its treatment
   * Known bleeding disorder (e.g., dysfibrinogenaemia, factor IX deficiency, haemophilia, Von Willebrand's disorder, Disseminated Intravascular Coagulation [DIC], fibrinogen deficiency, or other clotting factor deficiency)
10. Evidence at the time of Screening of significant renal or hepatic insufficiency (unless due to haemolysis, or leukaemic infiltration) as defined by any of the following local lab parameters:

    1. Calculated glomerular filtration rate (GFR; using the Cockcroft-Gault equation) < 40 mL/min or serum creatinine > 1.5 x the local upper limit of normal
    2. Aspartate transaminase (AST) or alanine aminotransferase (ALT) ≥ 2 x the local upper limit of normal
11. Current use of a prohibited medication (e.g., romiplostim) or expected to require any of these medications during treatment with the investigational drug.
12. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to IMG-7289 or LSD1 inhibitors (i.e., monoamine oxidase inhibitors; MAOIs) that contraindicates their participation.
13. Patients with impaired decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Hematologic Response Rates | 24 Weeks
  As evaluated by the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) and European Leukemia Net (ELN) response criteria.

SECONDARY OUTCOMES:
Incidence of Treatment-Related Toxicity | Up to 3 Years
  As evaluated by the treating physician using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Change in Total Symptom Score (TSS) as Measured by the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) | Baseline, Up to 3 Years
  As measured using the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) that includes 14 disease related symptoms each scored from 0 (absent) to 10 (worst imaginable).
Change in Mutational Allele Burden | Baseline, Up to 3 Years
  Evaluated via Next Generation Sequencing (NGS) molecular profiling from serum blood sample.
Change in Spleen Size in Centimeters | Baseline, Up to 3 Years
  Measured via physical examination and radiologic imaging measurement.
Change in Fibrosis Score | Baseline, Up to 3 Years
  Assessed using a slightly modified version of European Consensus Criteria for Grading Myelofibrosis from bone marrow/aspirate sample, as presented in Thiele et al, 2005. Myelofibrosis (MF) scores are graded on a four-point scale, from MF-0 to MF-3, grading the reticulin and collagen content of bone marrow, with MF-0 being the lowest and MF-3 the highest.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence J Bradley, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No